CLINICAL TRIAL: NCT00326690
Title: A Prospective, Randomized Trial Using a reproduciBLe volUmE-Measurement stratEGy in the surGical Reconstruction of the Ischemic Cardiomyopathic Heart
Brief Title: Study Tests Whether a Standardized LVR Performed With the Blue Egg Device Improves Cardiopulmonary Exercise Capacity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit and enroll patients
Sponsor: BioVentrix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioVentrix - Blue Egg Trial™
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Congestive Heart Failure; Ischemic Cardiomyopathy; Coronary Artery Disease; Myocardial Diseases
Keywords: Congestive Heart Failure; Coronary Artery Disease; Ischemic Cardiomyopathy; Idiopathic Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Cardiomyopathies

ARMS (2):
- treatment (Experimental)
  Interventions: Device: Blue Egg Device
- Control (No Intervention)

INTERVENTIONS:
Device: Blue Egg Device
  Arms: treatment

SUMMARY:
The purpose of the present prospective, randomized study is to investigate the clinical effectiveness of standardized left ventricular reconstruction surgery (LVR). In order to standardize the procedure, the operation will be performed with the Blue Egg, manufactured by BioVentrix, a subsidiary of CHF Technologies, Inc.

DETAILED DESCRIPTION:
The primary objective of this study is to test whether a standardized Left Ventricular Reconstruction (LVR) performed with the Blue Egg device improves cardiopulmonary exercise capacity in subjects with stable New York Heart Association (NYHA) Class III or IV heart failure due to ischemic cardiomyopathy with an akinetic or dyskinetic anterior wall. This shall be accomplished by comparing changes in cardiopulmonary exercise between a group of subjects treated with LVR and optimal medical therapy (Treatment) to a group treated with optimal medical therapy alone (Control).

Secondary objectives will examine the difference in heart failure symptoms between the two groups.

The primary hypothesis is that the average change in peak oxygen consumption (MVO2) observed in the treatment group from baseline to 6 months post surgery date is at least 1.2 ml O2/min/kg greater than the average change observed in the control group in the same time frame.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have symptomatic heart failure consistent with NYHA Class III or IV
* Have been treated, in the opinion of the Principal Investigator, for at least 12 weeks with an optimized pharmacological regimen, including no substantial dosage titration for the last 4 weeks. This will typically mean that the subject has had (unless intolerant) appropriate doses of angiotensin-converting enzyme (ACE) inhibitors, beta-blockers (β-blockers) and/or aldosterone inhibitors and diuretics.
* Have a dilated left ventricular (LV) with an LV end-systolic volume index (LVESVI) of 60 ml/m² and an akinetic or dyskinetic anterior wall
* Have an LV ejection fraction less than or equal to 35%
* Have an MVO2 of equal to or greater than 10, but equal to or less than 16 ml O2/min/kg
* Have demonstrated myocardial infarction without viability on a dobutamine stress echocardiogram in a region considered for surgery. Alternatively, have demonstrated the same physiological feature with gadolinium/magnetic resonance imaging (MRI) procedures or other sophisticated methodology for viability assessment.
* Agree to be compliant with the study protocol and willing and able to return for follow-up

Exclusion Criteria:

* Have had a myocardial infarction within 90 days of consent
* Be inotrope or intra-aortic balloon pump (IABP) dependent
* Require, in the judgment of the Principal Investigator, cardiac surgery that cannot be deferred for 6 months, such as subjects with:

  * left main coronary artery disease
  * intractable ventricular arrhythmias
  * Canadian Cardiovascular Society Angina Class III or IV symptoms
  * aortic stenosis or insufficiency requiring replacement
  * 3+ or 4+ mitral regurgitation
* Have any comorbid medical condition that is a contraindication to cardiac surgery (e.g., renal failure, coagulopathy, severe chronic obstructive pulmonary disease [COPD], cerebrovascular accident [CVA], prior stroke, known malignancy etc.)
* Have congestive heart failure (CHF) due to a cause other than ischemic cardiomyopathy
* Have a history of radiation therapy to the chest or mediastinum
* Have exercise tolerance limited by a condition other than heart failure
* Be unable to perform cardiopulmonary stress test
* Have a history of alcohol abuse, drug addiction, or other psychosocial condition that would preclude successful participation or realization of benefit from the trial in the opinion of the Principal Investigator.
* Be a female of child-bearing age who is pregnant or does not agree to use standard methods of birth control.
* Carry a diagnosis of an illness other than CHF with life expectancy less than 12 months.
* Participating in another trial (other than non-therapeutic or interventional observation) within the last 30 days or less than 60 days after completion of a heart failure drug trial.
* Biventricular pacemaker implantation and/or activation within the past 60 days
* Percutaneous coronary intervention (PCI) with coronary revascularization within the last 60 days.
* More than one prior sternotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
A change in peak oxygen consumption (MVO2) observed in the treatment group from baseline to 6 months post surgery date is at least 1.2 ml O2/min/kg greater than the average change observed in the control group in the same time frame. | 6 months

SECONDARY OUTCOMES:
Secondary objectives will examine the difference in heart failure symptoms between the two groups. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. Lazzara, MD, Principal Investigator — St. Joseph's Hospital; Ulrich Jorde, MD, Principal Investigator — New York College of Medicine; Francis Pagani, MD, Principal Investigator — University of Michigan; James D. Bergin, MD, Principal Investigator — University of Virginia College of Medicine; Howard J Eisen, MD, Principal Investigator — Drexel University College of Medicine; Ernst Schwarz, MD, Principal Investigator — Cedar Sinai Department of Cardiothoracic Surgery; Volkmar Falk, MD, Principal Investigator — Heart Center Leipzig; Mariell Jessup, MD, Principal Investigator — University of Pennsylvania; Erika Feller, MD, Principal Investigator — University of Maryland College of Medicine; Rosemary Peterson, MD, Principal Investigator — St. Joseph's Hospital - Tacoma, WA
Locations (10):
- United States (9):
  - Cedar Sinai Department of Cardiothoracic Surgery, Los Angeles, California
  - St. Joseph's Hospital, St. Petersburg, Florida
  - University of Maryland College of Medicine, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - NYU College of Medicine, New York, New York
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Virginia College of Medicine, Charlottesville, Virginia
  - St. Joseph's Hospital, Tacoma, Washington
- Heart Center Leipzig, Leipzig, Germany

REFERENCES:
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Athanasuleas CL, Stanley AW Jr, Buckberg GD, Dor V, DiDonato M, Blackstone EH. Surgical anterior ventricular endocardial restoration (SAVER) in the dilated remodeled ventricle after anterior myocardial infarction. RESTORE group. Reconstructive Endoventricular Surgery, returning Torsion Original Radius Elliptical Shape to the LV. J Am Coll Cardiol. 2001 Apr;37(5):1199-209. doi: 10.1016/s0735-1097(01)01119-6. PMID 11300423
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Cohn JN. The Vasodilator-Heart Failure Trials (V-HeFT). Mechanistic data from the VA Cooperative Studies. Introduction. Circulation. 1993 Jun;87(6 Suppl):VI1-4. No abstract available. PMID 8500232
- [Background] Hjalmarson A, Goldstein S, Fagerberg B, Wedel H, Waagstein F, Kjekshus J, Wikstrand J, El Allaf D, Vitovec J, Aldershvile J, Halinen M, Dietz R, Neuhaus KL, Janosi A, Thorgeirsson G, Dunselman PH, Gullestad L, Kuch J, Herlitz J, Rickenbacher P, Ball S, Gottlieb S, Deedwania P. Effects of controlled-release metoprolol on total mortality, hospitalizations, and well-being in patients with heart failure: the Metoprolol CR/XL Randomized Intervention Trial in congestive heart failure (MERIT-HF). MERIT-HF Study Group. JAMA. 2000 Mar 8;283(10):1295-302. doi: 10.1001/jama.283.10.1295. PMID 10714728
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Packer M, Coats AJ, Fowler MB, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Castaigne A, Roecker EB, Schultz MK, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival Study Group. Effect of carvedilol on survival in severe chronic heart failure. N Engl J Med. 2001 May 31;344(22):1651-8. doi: 10.1056/NEJM200105313442201. PMID 11386263
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Rose EA, Gelijns AC, Moskowitz AJ, Heitjan DF, Stevenson LW, Dembitsky W, Long JW, Ascheim DD, Tierney AR, Levitan RG, Watson JT, Meier P, Ronan NS, Shapiro PA, Lazar RM, Miller LW, Gupta L, Frazier OH, Desvigne-Nickens P, Oz MC, Poirier VL; Randomized Evaluation of Mechanical Assistance for the Treatment of Congestive Heart Failure (REMATCH) Study Group. Long-term use of a left ventricular assist device for end-stage heart failure. N Engl J Med. 2001 Nov 15;345(20):1435-43. doi: 10.1056/NEJMoa012175. PMID 11794191
- [Background] Starling RC, McCarthy PM, Buda T, Wong J, Goormastic M, Smedira NG, Thomas JD, Blackstone EH, Young JB. Results of partial left ventriculectomy for dilated cardiomyopathy: hemodynamic, clinical and echocardiographic observations. J Am Coll Cardiol. 2000 Dec;36(7):2098-103. doi: 10.1016/s0735-1097(00)01034-2. PMID 11127447
- [Background] Young JB, Abraham WT, Smith AL, Leon AR, Lieberman R, Wilkoff B, Canby RC, Schroeder JS, Liem LB, Hall S, Wheelan K; Multicenter InSync ICD Randomized Clinical Evaluation (MIRACLE ICD) Trial Investigators. Combined cardiac resynchronization and implantable cardioversion defibrillation in advanced chronic heart failure: the MIRACLE ICD Trial. JAMA. 2003 May 28;289(20):2685-94. doi: 10.1001/jama.289.20.2685. PMID 12771115